CLINICAL TRIAL: NCT05265832
Title: Identification of Factors That Influence the Corneal Endothelial Cell Loss During Phacoemulsification
Brief Title: Influencing Factors of the Corneal Endothelial Cell Loss
Acronym: PREDICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-04-CHRMT
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-11

CONDITIONS: Cataract
Keywords: Endothelial cell loss
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cataract surgery (Experimental): Phacoemulsification cataract surgery
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Endocapsular technique (Divide-and-conquer) and supracapsular technique (Subluxation) will be used equally.

SUMMARY:
This is a multi-center cohort study with prognostic aims to identify factors associated with endothelial cell loss during cataract surgery.

Patients will have their endothelial density measured by specular microscopy preoperatively, at 1 month and at 3 months after surgery. The rest of their management will be in line with standard practice.

DETAILED DESCRIPTION:
Cataract surgery is the most commonly performed surgical procedure worldwide. Postoperative visual function depends on implant into the crystalline lens, retinal lesion, corneal damage or glaucomatous damage. Moreover, preoperative corneal endothelial damage should be as low as possible to provide corneal transparency. Indeed, the endothelium plays important role in maintaining corneal transparency.

The loss rate of endothelial cell after cataract surgery ranges in the scientific literature from 8 to 15 %. Severe endothelial cell loss contributes to corneal edema. This edema resulting in a loss of visual acuity and may require corneal transplantation as a last resort.

Various studies describe some factors that affecting endothelial cell loss such as the cataract density, pupil abnormalities (small diameter), Advanced age or short axial length.

However, few studies have been demonstrated the link between endothelial cell loss and the volume of fluid used during the intervention or the use of intracamerular substances. This study wants to establish a correlation between endothelial cell loss and predictive factors. Thus, knowledge of these factors would have ensured a better control of endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery
* Visual acuity monoyer scale <8/10e (> +0.2 logMar)
* Nuclear, cortical and posterior subcapsular cataract with normal density to severe in the LOCSIII classification
* Covered by the social security scheme
* Have given their oral agreement

Exclusion Criteria:

* Corneal disease: keratitis, dystrophy or corneal degeneration
* Any disease of the anterior segment
* Low preoperative endothelial cell density <1000 c/mm²
* Pregnancy, lactation
* Risk factors for surgical per-operative complication
* Uncontrolled ocular pressure
* Combined surgery (cataract with corneal graft, cataract with glaucoma surgery, cataract with vitrectomy, ....)
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Postoperative endothelial cell loss | Month 3
  Difference in endothelial cell density between preoperative measurements and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Perone, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (2):
- France (2):
  - CHR Metz-Thionville/Hopital Mercy, Metz, Grand Est
  - CHR Metz-Thionville_Hopital Bel Air, Thionville, Grand Est